CLINICAL TRIAL: NCT04167696
Title: Open-label, Phase I, Multi-center Study to Determine in Relapsed/Refractory Acute Myeloid Leukemia or Myelodysplastic Syndrome Patients the Recommended Dose of CYAD-02 After a Non-myeloablative Preconditioning Chemotherapy Followed by a Potential Consolidation Cycle
Brief Title: Study in Relapsed/Refractory Acute Myeloid Leukemia or Myelodysplastic Syndrome Patients to Determine the Recommended Dose of CYAD-02
Acronym: CYCLE-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Celyad Oncology SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CYAD-02-001
Record Dates: First submitted 2019-11-12; First posted 2019-11-19 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Cyclophosphamide; fludarabine phosphate; fludarabine

STUDY DESIGN:
Intervention Model Description: Dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation Dose Level 1 (Experimental): in case of no dose limiting toxicity (DLT) and no replacement of patients, 3 consecutive patients at the dose of 1x10e8 of CYAD-02 per infusion post preconditioning non-myeloablative chemotherapy according to a 3+3 study design.
  The preconditioning therapy consists of 3 consecutive days of cyclophosphamide (300 mg/m²/day) and fludarabine (30 mg/m²/day), two days before the CYAD-02 infusion.
  In case of no progression at D22, the patient is eligible to receive a consolidation cycle of 3 additional CYAD-02 infusion at the same dose level, without prior preconditioning chemotherapy.
  Interventions: Biological: CYAD-02; Drug: ENDOXAN; Drug: Fludara
- Dose Escalation Dose Level 2 (Experimental): in case of no dose limiting toxicity (DLT) and no replacement of patients,3 consecutive patients at the dose of 3x10e8 of CYAD-02 per infusion post preconditioning non-myeloablative chemotherapy according to a 3+3 study design.
  The preconditioning therapy consists of 3 consecutive days of cyclophosphamide (300 mg/m²/day) and fludarabine (30 mg/m²/day), two days before the CYAD-02 infusion.
  In case of no progression at D22, the patient is eligible to receive a consolidation cycle of 3 additional CYAD-02 infusion at the same dose level, without prior preconditioning chemotherapy.
  Interventions: Biological: CYAD-02; Drug: ENDOXAN; Drug: Fludara
- Dose Escalation Dose Level 3 (Experimental): in case of no dose limiting toxicity (DLT) and no replacement of patients,3 consecutive patients at the dose of 1x10e9 of CYAD-02 per infusion post preconditioning non-myeloablative chemotherapy according to a 3+3 study design.
  The preconditioning therapy consists of 3 consecutive days of cyclophosphamide (300 mg/m²/day) and fludarabine (30 mg/m²/day), two days before the CYAD-02 infusion.
  In case of no progression at D22, the patient is eligible to receive a consolidation cycle of 3 additional CYAD-02 infusion at the same dose level, without prior preconditioning chemotherapy.
  Interventions: Biological: CYAD-02; Drug: ENDOXAN; Drug: Fludara

INTERVENTIONS:
Biological: CYAD-02 — CYAD-02 is a Chimeric Antigen Receptor-T (CAR-T) administered after CYFLU.
Drug: ENDOXAN — administered as preconditioning chemotherapy
  Other Names: cyclophosphamide
Drug: Fludara — administered as preconditioning chemotherapy
  Other Names: fludarabine

SUMMARY:
An open-label, phase I, multi-center study to determine in relapsed/refractory (r/r) acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) patients the recommended dose of CYAD-02 after a non-myeloablative preconditioning chemotherapy followed by a potential CYAD-02 consolidation cycle for non-progressive patient. A maximum of 27 r/r AML/MDS patients will be evaluated in this study in case of no dose limiting toxicity (DLT) and no replacement of patients.

DETAILED DESCRIPTION:
This open-label phase I, multi-center study aims to determine in relapsed/refractory acute myeloid leukemia or myelodysplastic syndrome patients the recommended dose of CYAD-02 after a non-myeloablative preconditioning chemotherapy followed by a potential CYAD-02 consolidation cycle for non-progressive patients.

During dose escalation, three prespecified dose-levels of CYAD-02 will be evaluated in three cohorts. Patient enrollment during dose-escalation will be staggered according to the Fibonacci 3+3 design and extension of cohorts II and III will be done in parallel. The first CYAD-02 infusion will be administered after prior non-myeloablative preconditioning chemotherapy (CYFLU) administered on three consecutive days.

Non-progressive patients meeting the criteria specified below may receive a consolidation cycle with three additional CYAD-02 infusions at a 2-week interval without prior preconditioning.

For all patients who received at least one CYAD-02 infusion, the overall study duration will be approximately 15 years.

ELIGIBILITY:
Inclusion Criteria (main):

* The patient must not be eligible for standard of care therapy and have one of the following hematological malignancy:

  1. A confirmed relapsed or refractory acute AML (i.e. ≥ 5% blasts in bone marrow or in peripheral blood) with revised European LeukemiaNet (ELN) 2017 risk stratification for favorable, intermediate or adverse groups, after at least one prior therapy defined as either

     * Recurrence of disease after a first complete remission and not eligible for a second course of induction therapy, or
     * Recurrence of disease after a second complete remission, or
     * Failure to achieve a Complete Response after induction chemotherapy.
  2. A confirmed MDS as defined by revised International Prognostic Scoring System criteria for intermediate, high-risk or very high-risk disease or MDS with Tumor Protein 53 mutation as detected by next-generation sequencing, after failure of prior treatment with at least 4 cycles of azacitidine or decitabine defined as:

     * No response to treatment,
     * Loss of response at any time point, or
     * Intolerance to therapy.
* The patient must have evaluable disease as defined by:

  * Revised Recommendations of the International Working Group (IWG) for Diagnosis, Standardization of Response Criteria for AML patients,
  * IWG 2006 Uniform Response Criteria for patients with MDS.
* The absolute peripheral blast count should be < 15,000/L.
* The patient must have adequate hepatic and renal functions, as assessed by standard laboratory criteria.
* The patient must have a left ventricular ejection fraction of ≥ 40 %, as determined by echocardiography or a multigated acquisition scan.
* The patient must have a Forced Expiratory Volume (FEV) in the first second /Forced Vital Capacity = 0.7 with FEV-1 at 50 % predicted (GOLD 1 or 2 severity) as determined by spirometry

Exclusion Criteria (main):

* Patients with a confirmed or history of tumor involvement in the central nervous system
* Patients who have received any cancer therapy with therapeutic intent (investigational agent or not)
* Patients with any positive serology test results at baseline
* Patients who plan to receive, are concurrently receiving or have received any investigational agent within 3 weeks before the planned day for the first CYAD-02 infusion
* Patients with uncontrolled intercurrent illness or serious uncontrolled medical disorder
* Patients with significant coagulation disorder or who are receiving treatment with warfarin derivatives, heparin or direct oral anticoagulants
* Patients who have active infections
* Patients with documented history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis and/or active or acute exacerbation of chronic obstructive pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2035-02 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicities as defined per protocol in order to define the final recommended dose. | from start the first infusion of CYAD-02 (Day1) up to Day36.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - University of Kansas Cancer Center, Fairway, Kansas
- Belgium (3):
  - Uz Leuven, Leuven
  - Chu Liege, Liège
  - AZ DELTA, Roeselare

IPD SHARING:
Plan to Share IPD: No